CLINICAL TRIAL: NCT00387127
Title: A Randomized, Double-blind, Placebo Controlled, Multicentre, Phase II Study of Oral Lapatinib in Combination With Concurrent Radiotherapy and Cisplatin Versus Radiotherapy and Cisplatin Alone, in Subjects With Stage III, IVA, B Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Lapatinib Versus Placebo Given Concurrently With Cisplatin And Radiotherapy In Patients With Unresected Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGF105884
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms, Head and Neck
Keywords: Neck Cancer; Locally advanced head and neck cancer; locally advanced; Head and Neck cancer; lapatinib; EGFR/ErbB2 inhibitor; Head Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Lapatinib; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lapatinib (Experimental): 1500mg lapatinib orally daily
  Interventions: Drug: Lapatinib oral tablets; Drug: radiotherapy; Drug: cisplatin chemotherapy
- Placebo (Placebo Comparator): orally daily
  Interventions: Drug: Lapatinib oral tablets; Drug: radiotherapy; Drug: cisplatin chemotherapy

INTERVENTIONS:
Drug: Lapatinib oral tablets — Lapatinib is administered orally once daily.
Drug: radiotherapy — Radiotherapy is given either as conventional fractionation using Two-dimensional (2D) or conformal techniques, or as Intensity Modulated Radiation Therapy (IMRT). Radiation therapy will be standardised throughout the study. Radiation therapy is given only once daily, with a dose/fraction not exceeding 2.5Gy, to a total dose of 65 Gy (IMRT) or 70 Gy (2D or 3D RT) to the gross site of disease .
Drug: cisplatin chemotherapy — Cisplatin is administered intravenously at a dose of 100mg/m2 on days 1, 22 and 43 of radiotherapy (approximately Study Days 8, 29 and 50).
  Other Names: radiotherapy; Lapatinib oral tablets

SUMMARY:
This is a phase II study comparing the effects of lapatinib versus placebo when administered concurrently with cisplatin and radiotherapy followed by 1 year monotherapy with lapatinib or placebo. The study is designed to evaluate and compare the two treatment groups with respect to complete response rate at 6 months following chemoradiation completion.

ELIGIBILITY:
Inclusion criteria:

* Willing and able to sign a written informed consent;
* Histologically confirmed diagnosis of SCCHN of one or more of the following sites:

oral cavity, oropharynx, hypopharynx and larynx;

Multiple primary tumours will:

Have to be histologically proven; Have to be anatomically distant and surrounded by normal tissue; Exclude distant metastasis.

* Prior to enrolment subjects must have ErbB1 over-expression determined by immunohistochemistry (IHC) 3+ as assessed by a central laboratory;
* Subjects with stage III and IVA/IVB disease, who are to receive cisplatin chemotherapy and radiation therapy as primary treatment (total dose 65 - 70 Gy); Subjects with any Tis, T1 or T2 disease regardless of N stage, are excluded. Subjects with distant metastases, ie Stage IVC, are excluded.
* Willing and able to have a tumour biopsy taken at screening; For patients who have had prior tumour biopsy, an adequate archived specimen must be available.
* Male or female ≥18 years of age;

Criteria for female subjects or female partners of male subjects:

Non-child-bearing potential (i.e., women with functioning ovaries who have a GM2005/00448/00 CONFIDENTIAL EGF105884 22 current documented tubal ligation or hysterectomy, or women who are postmenopausal); Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at screening and agree to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or Consistent and correct use of one of the following acceptable methods of birth control: male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; implants of levonorgestrel; injectable progestogen; any intrauterine device (IUD) with a documented failure rate of less than

1% per year; oral contraceptives (either combined or progestogen only); or barrier methods, including diaphragm or condom with a spermicide.

* ECOG performance status 0, 1 or 2;
* Subjects must have adequate haematological, renal and hepatic function; Calculated creatinine clearance ≥50 ml/min as determined by the modified method of Cockcroft and Gault or by the EDTA method. Absolute neutrophil count ≥1,500/μl, platelets ≥100,000/μl. Haemoglobin ≥9gm/dL (5mmol/L). Aspartate (AST) and alanine transaminase (ALT) less than 4 times the upper limit of the normal range (ULN). Total bilirubin ≤2.0 mg/dL.
* Left ventricular ejection fraction (LVEF) within the institutional normal ranges as measured by echocardiogram (ECHO) or Multigated Acquisition (MUGA) scan;
* Able to swallow tablets whole or swallow a suspension of tablets dissolved in water at study inclusion; The use and timing of feeding tube is optional. If necessary, the suspension may be administered via percutaneous endoscopic gastrostomy (PEG), percutaneous jejunostomy tube (J- Tube), or a nasogastric tube (NG or Dobhoff type tube).
* Life expectancy of at least 6 months in the best judgment of the investigator.

Exclusion criteria:

* Nasopharyngeal, paranasal sinuses or nasal cavity tumours;
* Any prior or current treatment for invasive head and neck cancer of any kind. This will include but is not limited to: prior tyrosine kinase inhibitors, prior neoadjuvant therapy, prior surgical resection, or use of any investigational agent;
* Concurrent use of CYP3A4 inducers or inhibitors. A standard 3-day course of dexamethasone for the prevention of cisplatin-induced nausea and vomiting is permitted;
* Subjects with known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure;
* History of another malignancy within the last 5 years, with the exception of completely resected basal or squamous cell skin cancer, or successfully treated in-situ carcinoma. History of non-invasive lesion or in-situ carcinoma, including in the head and neck region that was successfully treated with surgery, photodynamics or laser, will be permitted;
* Peripheral neuropathy ≥ grade 2;
* Pregnant or lactating females (female subjects of child-bearing potential will undertake pregnancy testing at screening and during study completion/withdrawal visits);
* Malabsorption syndrome, disease significantly affecting GI function, that could affect absorption of lapatinib;
* History of allergic reactions to appropriate antiemetics (e.g. 5-HT3 antagonists) to be administered with platinum chemotherapy;
* The investigator considers the subject unfit for the study as a result of the medical interview, physical examinations, or screening investigations;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (3):
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
- Canada (3):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- France (5):
  - GSK Investigational Site, Lens
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
- India (3):
  - GSK Investigational Site, Ahemdabad
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Thiruvananthapuram
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leiden
- GSK Investigational Site, Lima, Lima Province, Peru
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- United Kingdom (7):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Background] Harrington K, Berrier A, Robinson M, Remenar E, Housset M, de Mendoza FH, Fayette J, Mehanna H, El-Hariry I, Compton N, Franklin N, Biswas-Baldwin N, Lau M, Legenne P, Kumar R. Randomised Phase II study of oral lapatinib combined with chemoradiotherapy in patients with advanced squamous cell carcinoma of the head and neck: rationale for future randomised trials in human papilloma virus-negative disease. Eur J Cancer. 2013 May;49(7):1609-18. doi: 10.1016/j.ejca.2012.11.023. Epub 2012 Dec 19. PMID 23265705
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiotherapy + Placebo, Followed by Placebo: Participants received radiotherapy once daily (OD), with a dose/fraction <2.5 Gray (Gy) to a total dose of 70 Gy (using two-dimensional [2D] or 3D techniques) or 65 Gy (using Intensity Modulated Radiation Therapy [IMRT]) to the gross site of disease. Concurrent chemotherapy of cisplatin 100 milligrams per meters squared (mg/m^2) was administered intravenously (IV) on Days 1, 22, and 43 of the course of radiotherapy (Study Days 8, 29, and 50). Matching placebo administration commenced 1 week (or less than or equal to 3 days) prior to the concurrent administration with chemoradiation for a duration of up to 6 to 7 weeks. After the completion of chemoradiotherapy, placebo monotherapy was administered until disease progression or withdrawal.
- Chemoradiotherapy + Lapatinib, Followed by Lapatinib: Participants received radiotherapy once daily (OD), with a dose/fraction <2.5 Gy to a total dose of 70 Gy (using 2D or 3D techniques) or 65 Gy (using IMRT) to the gross site of disease. Concurrent chemotherapy of cisplatin 100 mg/m^2 was administered IV on Days 1, 22, and 43 of the course of radiotherapy (Study Days 8, 29, and 50). Lapatinib 1500 mg OD administration commenced 1 week (or less than or equal to 3 days) prior to the concurrent administration with chemoradiation for a duration of up to 6 to 7 weeks. After the completion of chemoradiotherapy, lapatinib 1500 mg OD monotherapy was administered until disease progression or withdrawal.
Period: Overall Study
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Started | 33 | 34
Completed | 0 | 0
Not Completed | 33 | 34
Not completed — Lost to Follow-up | 0 | 4
Not completed — Death | 16 | 16
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Required by Protocol Amendment #4 | 12 | 10
Not completed — Serious Adverse Event | 1 | 1
Not completed — Sponsor Unblinded | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (6.61) | 55.8 (5.73) | 56.1 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 31 | 29 | 60
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 1 | 1
  American Indian or Alaska Native | 2 | 2 | 4
  Asian - Central/South Asian Heritage | 3 | 6 | 9
  Asian - South East Asian Heritage | 2 | 1 | 3
  White - White/Caucasian/European Heritage | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Complete Response (CR), as Assessed by Independent Radiological Review
Description: Participants with CR are defined as those who achieved a complete tumor response at 6 months after the completion of the chemoradiation treatment (CRT), as assessed by independent radiological review. Tumor response was assessed using modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Per RECIST, CR is defined as the disappearance of all target and non-target lesions. Data are based on Week 24 scans from participants receiving study treatment at that time and on those in follow-up.
Time Frame: From the date of randomization until 6 months post chemoradiation treatment, assessed for a median time of 13 months
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to study treatment, regardless of whether they actually received study medication
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants | 12 | 18
Statistical Analysis 1: Comparison: Chemoradiotherapy + Placebo, Followed by Placebo vs Chemoradiotherapy + Lapatinib, Followed by Lapatinib; Test type: Superiority or Other; p = 0.3658, Fisher Exact — From exact test that common odds ratio equals 1; Difference in percentage of par. with CR = 10.7, 95% CI 2-sided [-13.4 to 37.3] — Complete response was defined as the percentage of participants achieving a CR as determined by an independent radiological review

2. Secondary Outcome: Number of Participants With CR, as Assessed by the Investigator
Description: Participants with CR are defined as those who achieved a complete tumor response at 6 months after the completion of the CRT, as determined by the investigator. Tumor response was assessed using modified RECIST criteria. Per RECIST, CR is defined as the disappearance of all target and non-target lesions. Data are based on Week 24 scans from participants receiving study treatment at that time and on those in follow-up.
Time Frame: From the date of randomization until 6 months post chemoradiation treatment, assessed after a median time of 13 months of follow-up
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants | 7 | 17
Statistical Analysis 1: Comparison: Chemoradiotherapy + Placebo, Followed by Placebo vs Chemoradiotherapy + Lapatinib, Followed by Lapatinib; Test type: Superiority or Other; p = 0.0130, Fisher Exact — From exact test that common odds ratio equals 1; Difference in percentage of par. with CR = 28.8, 95% CI 2-sided [5.7 to 53.6] — Complete response was defined as the percentage of participants achieving a CR as determined by the investigator

3. Secondary Outcome: Progression-Free Survival (PFS), as Assessed by the Investigator
Description: PFS=the time from randomization until the earliest date of disease progression or death due to any cause, if sooner. Per RECIST, progressive disease=a >=20% increase in the sum of the longest diameter of target lesions (TLs), or the appearance of >=1 new L, symptomatic progression and/or unequivocal progression of existing non-TLs. For participants who did not progress or die at the time of reporting (data cut-off 1-Aug-2014), PFS data were censored at the time of the last investigator assessed radiological scan preceding the initiation of any alternative anti-cancer therapy.
Time Frame: From the date of randomization until the date of disease progression or death due to any cause, assessed after a median of 22 months of follow-up
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Months | 12.1 [7.3 to NA] — There were too few events to allow for the calculation of the upper limit of the confidence interval. | 20.4 [10.8 to NA] — There were too few events to allow for the calculation of the upper limit of the confidence interval.

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death due to any cause. Time to death (data cut-off 1-Aug-2014) was censored at the time of last contact for participants who did not die.
Time Frame: From the date of randomization until the date of death due to any cause, assessed after a median of 30.9 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Months | 23.0 [14.2 to NA] — There were too few events to allow for the calculation of the upper limit of the confidence interval. | 48.4 [18.8 to NA] — There were too few events to allow for the calculation of the upper limit of the confidence interval.

5. Secondary Outcome: Number of Participants Who Died Due to Progressive Disease
Description: The number of participants who died due to progressive disease (a >=20% increase in the sum of the longest diameter of target lesions, or the appearance of >=1 new lesion, symptomatic progression and/or unequivocal progression of existing non-target lesions), or died due to head and neck cancer without evidence of disease progression, after randomization in the study is presented, using a data cut of 1 August 2014.
Time Frame: From the date of randomization until the date of death due to disease under study, assessed after a median of 30.9 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants | 11 | 8

6. Secondary Outcome: Disease-specific Survival
Description: Disease-specific survival is defined as the time from randomization until death due to head and neck cancer.
Time Frame: From the date of randomization until the date of death due to disease, assessed after a median of 13 months of follow-up
Population: ITT Population. For participants who did not die, time to death was censored at the time of last contact.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Months | NA [15.6 to NA] — The cumulative incidence in the placebo arm remained lower than 50%, so the median and upper quartile were not observed. | NA [NA to NA] — The cumulative incidence remained lower than 25% in the lapatinib arm, so neither the median nor the inter-quartile range were observed.

7. Secondary Outcome: Number of Participants With Loco-regional Recurrence of Initial Disease
Description: Participants with loco-regional recurrence were those who had progression of disease in the T and N sites. Per the Tumor, Node, and Metastases (TNM) staging of tumors: T describes the size of the tumor and whether it has invaded nearby tissue, and N describes regional lymph nodes that are involved. If a participant had progression in the T or N sites, then the participant was counted as having had an event of interest.
Time Frame: From the date of randomization until progression in the T or N site or death due to any cause, assessed after a median of 30.9 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants | 7 | 4

8. Secondary Outcome: Loco-regional Control
Description: Loco-regional control is defined as the time from the date of randomization until progression in the T or N site. Participants who died or had secondary primary malignancies in the head and neck region outside of the T and N site or distant metastasis were not counted as an event and were instead treated as competing risks. Per the TNM staging of tumors: T describes the size of the tumor and whether it has invaded nearby tissue, and N describes regional lymph nodes that are involved. Due to the minimal events reported (data cut-off 30-Sep-2010), valid analysis could not be performed for loco-regional control rate.
Time Frame: as for outcome 7
Population: ITT Population
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Distant Recurrence of Initial Disease
Description: Participants were analyzed for the occurrence of distant metastasis (spread of a disease from one organ or part to another non-adjacent organ or part) after randomization in the study until data cut-off date 1-Aug-2014. Participants who died or had recurrence of disease in the T or N sites or secondary primary malignancies in the head and neck region outside of the original T and N site were not counted as an event and were instead treated as competing risks.
Time Frame: From the date of randomization until the first occurrence of distant metastasis, assessed after a median of 30.9 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants | 5 | 8

10. Secondary Outcome: Distant Relapse
Description: Distant relapse is defined as the time from the date of randomization until the first occurrence of distant metastasis (spread of a disease from one organ or part to another non-adjacent organ of part). Participants who died or had recurrence of disease in the T or N sites or secondary primary malignancies in the head and neck region outside of the original T and N site were not counted as an event and were instead treated as competing risks.
Time Frame: From the date of randomization until the first occurrence of distant metastasis, assessed after a median of 30.9 months
Population: ITT Population. If a participant had a distant metastasis and then died, then the participant was counted as having had an event of interest.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Months | NA [NA to NA] — The cumulative incidence remained below 25% in the placebo arm, so neither the median nor the inter-quartile range were observed. | NA [56.8 to NA] — The cumulative incidence in the lapatinib arm did not reach 50% (most participants had not relapsed), so the median and the upper limit of the interquartile range were not observed.

11. Secondary Outcome: Number of Participants With Overall Response (OR), as Assessed by the Investigator
Description: Participants with OR were those who achieved either a CR or partial response (PR) from the assessment of overall tumor response at 6 months (24 weeks) following completion of CRT (data cut-off 30-Sep-2010). Per RECIST, CR is defined as the disappearance of all target and non-target lesions; PR is defined as at least a 30% decrease in the sum of the long diameter (LD) of target lesions, taking as a reference, the baseline sum LD. Data are based on Week 24 scans from participants receiving study treatment at that time point.
Time Frame: From the date of randomization until 6 months post chemoradiation treatment, assessed for a median of 13 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants | 15 | 21
Statistical Analysis 1: Comparison: Chemoradiotherapy + Placebo, Followed by Placebo vs Chemoradiotherapy + Lapatinib, Followed by Lapatinib; Test type: Superiority or Other; p = 0.1969, Fisher Exact — From exact test that common odds ratio equals 1; Difference in overall response rate = 16.3, 95% CI 2-sided [-8.6 to 42.1] — Overall response was defined as the percentage of participants achieving a PR or CR as determined by the investigator

12. Secondary Outcome: Number of Participants Positive and Negative for the Expression of Biomarkers in Tumor Tissue: Human Epidermal Growth Factor Receptor (HER)-1, HER2, HER3, HER4, P16, and Transforming Growth Factor (TGF-alpha)
Description: Paraffin-embedded tissue block (or sections) from archived tumor tissue sample, if available (from time of original diagnosis) or fresh tumor tissue, was sent for testing to determine intra-tumoral biomarker expression by immunohistochemistry (IHC) or fluorescent in situ hybridization (FISH) assay. Stained tumor slides or tissue micro arrays (TMAs) were scored by a pathologist from 0 (no expression) to 3+ (high expression). An expression level of >=2+ was considered positive.
Time Frame: Up to 28 days prior to the date of the first dose of lapatinib/placebo start
Population: ITT Population. Only those participants who had sufficient tumor sample for testing were analyzed.
Measure: Number; unit: Participants
Groups:
- Chemoradiotherapy + Lapatinib, Followed by Lapatinib: Participants received radiotherapy once daily (OD), with a dose/fraction <2.5 Gy to a total dose of 70Gy (using 2D or 3D techniques) or 65 Gy (using IMRT) to the gross site of disease. Concurrent chemotherapy of cisplatin 100 mg/m^2 was administered IV on Days 1, 22, and 43 of the course of radiotherapy (Study Days 8, 29, and 50). Lapatinib 1500 mg OD administration commenced 1 week (or less than or equal to 3 days) prior to the concurrent administration with chemoradiation for a duration of up to 6 to 7 weeks. After the completion of chemoradiotherapy, lapatinib 1500 mg OD monotherapy was administered until disease progression or withdrawal.
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 30 | 27
Participants
  HER1, Positive, n=27, 24 | 27 | 19
  HER1, Negative, n=27, 24 | 0 | 5
  HER2, Positive, n=26, 25 | 3 | 0
  HER2, Negative, n=26, 25 | 23 | 24
  HER2, Missing, n=26, 25 | 0 | 1
  HER3, Positive, n=27, 22 | 8 | 5
  HER3, Negative, n=27, 22 | 18 | 16
  HER3, Missing, n=27, 22 | 1 | 1
  HER4, Positive, n=26, 25 | 0 | 0
  HER4, Negative, n=26, 25 | 26 | 24
  HER4, Missing, n=26, 25 | 0 | 1
  P16 Positive, n=23, 23 | 3 | 4
  P16, Negative, n=23, 23 | 20 | 19
  TGF-alpha, Positive, n=24, 25 | 7 | 4
  TGF-alpha, Negative, n=24, 25 | 17 | 20
  TGF-alpha, Missing, n=24, 25 | 0 | 1

13. Secondary Outcome: Plasma Proteome Analysis
Description: Proteomic analyses of blood plasma samples were to be conducted to identify any changes in the proteome profile that could be related to the treatment response. Examination of pre-dosing (screening) plasma protein profiles could uncover novel blood-borne protein candidate biomarkers/profiles, which could be used to predict drug response.
Time Frame: From up to 28 days prior to the first dose of lapatinib/placebo start to 8 weeks after the first dose
Population: ITT Population. Plasma proteome data have not been analyzed (tested); thus, data are not available to disclose. Based on the negative outcome of Study EGF102988 (NCT00424255), no suitable analyses have been proposed for this small sample size.
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Analysis of Deoxyribonucleic Acid (DNA) and Ribonucleic Acid (RNA) From Tumor Samples
Description: No analysis was performed for tumor sample RNA/DNA.
Time Frame: Screening
Population: ITT Population. DNA/RNA from tumors has not been analyzed (tested); therefore, data are not available. No suitable analyses of DNA/RNA have been proposed for this small sample size of tumor samples.
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants Negative and Positive for Human Papilloma Virus (HPV) Infection, as Determined From Tumor Samples
Description: Analysis was performed for HPV infection analysis from the tumor biopsy samples obtained during the Screening period. p16 was used as a marker for HPV; thus, "negative" participants did not have the p16 marker.
Time Frame: Up to 28 days prior to the first dose of lapatinib/placebo
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants
  Negative | 20 | 19
  Positive | 3 | 4
  Unknown | 10 | 11

16. Secondary Outcome: Number of Participants Positive and Negative for Biomarker HER1/ErbB1 Categorized in the Indicated Independent Review Panel-assessed Tumor Responses by Expression of Biomarkers From Tumor Tissue: Sensitivity Analysis - 0 Versus (1, 2, 3)
Description: Tumor tissue (fresh or archived) was sent to a central laboratory for biomarker HER1/ErbB1 and tumor genetics analysis up to 1 week after randomization. Per RECIST: CR, disappearance of all lesions; PR, a >=30% decrease in the sum of the longest dimensions (LD) of the target lesions (TLs) taking as a reference the baseline sum LD; Progressive disease (PD), a >=20% increase in the sum of the LD of TLs, or the appearance of >=1 new lesion; Stable Disease (SD), neither PR nor PD, persistence of >=1 non-TL. 0=negative; 1, 2, 3=positive (increasing level of biomarker expression).
Time Frame: From the date of randomization until 6 months post chemoradiation treatment, assessed for up to 24 weeks
Population: ITT Population. Participants assessed for HER1/ ErbB1 expression were analyzed.
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 27 | 24
Participants
  Negative, CR | 0 | 0
  Negative, PR | 0 | 0
  Negative, SD | 0 | 0
  Negative, PD (Week 24) | 0 | 0
  Negative, PD or Death (prior to Week 24) | 0 | 0
  Negative, Not Evaluable | 0 | 0
  Negative, Unknown | 0 | 0
  Positive, CR | 9 | 14
  Positive, PR | 4 | 3
  Positive, SD | 0 | 0
  Positive, PD (Week 24) | 4 | 1
  Positive, PD or Death (prior to Week 24) | 5 | 4
  Positive, Not Evaluable | 1 | 0
  Positive, Unknown | 4 | 2

17. Secondary Outcome: Number of Participants Positive and Negative for Biomarker HER1/ErbB1 Categorized in the Indicated Independent Review Panel-assessed Tumor Responses by Expression of Biomarkers From Tumor Tissues: Sensitivity Analysis - 0, 1, 2 Versus 3
Description: as for outcome 16
Time Frame: From the date of randomization until 6 months post chemoradiation treatment, assessed for up to 24 weeks
Population: ITT Population. Participants assessed for HER1/ ErbB1 expression were analyzed.
Measure: Number; unit: Participants
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 33 | 34
Participants
  Negative, CR | 5 | 9
  Negative, PR | 2 | 2
  Negative, SD | 0 | 0
  Negative, PD (Week 24) | 1 | 0
  Negative, PD or Death (prior to Week 24) | 2 | 4
  Negative, Not Evaluable | 0 | 0
  Negative, Unknown | 1 | 1
  Positive, CR | 4 | 5
  Positive, PR | 2 | 1
  Positive, SD | 0 | 0
  Positive, PD (Week 24) | 3 | 1
  Positive, PD or Death (prior to Week 24) | 3 | 0
  Positive, Not Evaluable | 1 | 0
  Positive, Unknown | 3 | 1

18. Other Pre Specified Outcome: Number of Participants Classified as Responders, as Per Volumetric Tumor Response
Description: No analysis was not performed.
Time Frame: From the date of randomization until 6 months post chemoradiation treatment, assessed for a median of 13 months
Population: ITT Population. A formal analysis of this outcome measure was never performed; thus data are not available and cannot be reported.
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data are presented as of the cut-off date of 1-August-2014.
Description: Data are presented for the Safety Population (SP)=participants (par.) who were randomized and took >=1 dose of study medication (SM). One par. randomized to placebo received lapatinib in error and was assigned to the lapatinib arm in the SP. One par. randomized to placebo withdrew from the study prior to receiving SM and was not included in the SP.
Groups:
- Chemoradiotherapy + Placebo, Followed by Placebo: Participants received radiotherapy once daily (OD), with a dose/fraction less than 2.5 Gray (Gy) to a total dose of 70 Gy (using two-dimensional [2D] or 3D techniques) or 65 Gy (using Intensity Modulated Radiation Therapy [IMRT]) to the gross site of disease. Concurrent chemotherapy of cisplatin 100 milligrams per meters squared (mg/m^2) was administered intravenously (IV) on Days 1, 22, and 43 of the course of radiotherapy (Study Days 8, 29, and 50). Matching placebo administration commenced 1 week (or less than or equal to 3 days) prior to the concurrent administration with chemoradiation for a duration of up to 6 to 7 weeks. After the completion of chemoradiotherapy, placebo monotherapy was administered until disease progression or withdrawal.
- Chemoradiotherapy + Lapatinib, Followed by Lapatinib: Participants received radiotherapy once daily (OD), with a dose/fraction less than 2.5 Gy to a total dose of 70 Gy (using 2D or 3D techniques) or 65 Gy (using IMRT) to the gross site of disease. Concurrent chemotherapy of cisplatin 100 mg/m^2 was administered IV on Days 1, 22, and 43 of the course of radiotherapy (Study Days 8, 29, and 50). Lapatinib 1500 mg OD administration commenced 1 week (or less than or equal to 3 days) prior to the concurrent administration with chemoradiation for a duration of up to 6 to 7 weeks. After the completion of chemoradiotherapy, lapatinib 1500 mg OD monotherapy was administered until disease progression or withdrawal.
Arm/Group | Chemoradiotherapy + Placebo, Followed by Placebo | Chemoradiotherapy + Lapatinib, Followed by Lapatinib
Serious Adverse Events (participants affected / at risk) | 18/31 | 22/35
Other Adverse Events (participants affected / at risk) | 31/31 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiotherapy + Placebo, Followed by Placebo (N=31) | Chemoradiotherapy + Lapatinib, Followed by Lapatinib (N=35)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 2
Mucosal Inflammation (General disorders) | 1 | 3
Pneumonia (Infections and infestations) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Hemorrhage (Vascular disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal Tubular Disorder (Renal and urinary disorders) | 0 | 2
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Weight Decreased (Investigations) | 2 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Creatinine Renal Clearance Decreased (Investigations) | 0 | 1
Death (General disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Ejection Fraction Decreased (Investigations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Gastrostomy Failure (Injury, poisoning and procedural complications) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Localised Edema (General disorders) | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mouth Hemorrhage (Gastrointestinal disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Parotid Gland Inflammation (Gastrointestinal disorders) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pharyngeal Ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Soft Tissue Inflammation (General disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiotherapy + Placebo, Followed by Placebo (N=31) | Chemoradiotherapy + Lapatinib, Followed by Lapatinib (N=35)
Nausea (Gastrointestinal disorders) | 17 | 22
Mucosal Inflammation (General disorders) | 14 | 14
Dry Mouth (Gastrointestinal disorders) | 13 | 15
Vomiting (Gastrointestinal disorders) | 10 | 14
Constipation (Gastrointestinal disorders) | 13 | 9
Neutropenia (Blood and lymphatic system disorders) | 13 | 7
Weight Decreased (Investigations) | 12 | 11
Anemia (Blood and lymphatic system disorders) | 11 | 9
Diarrhea (Gastrointestinal disorders) | 2 | 18
Dysphagia (Gastrointestinal disorders) | 11 | 10
Asthenia (General disorders) | 14 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Pyrexia (General disorders) | 6 | 11
Odynophagia (Gastrointestinal disorders) | 9 | 7
Oral Pain (Gastrointestinal disorders) | 8 | 7
Radiation Skin Injury (Injury, poisoning and procedural complications) | 9 | 5
Dysgeusia (Nervous system disorders) | 8 | 5
Leukopenia (Blood and lymphatic system disorders) | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 8 | 17
Skin Reaction (Skin and subcutaneous tissue disorders) | 5 | 8
Headache (Nervous system disorders) | 6 | 6
Stomatitis (Gastrointestinal disorders) | 6 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Hemoglobin Decreased (Investigations) | 7 | 7
Hypokalemia (Metabolism and nutrition disorders) | 4 | 7
Localized Edema (General disorders) | 7 | 4
Creatinine Renal Clearance Decreased (Investigations) | 4 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Oral Candidiasis (Infections and infestations) | 6 | 4
Anxiety (Psychiatric disorders) | 4 | 5
Blood Creatinine Increased (Investigations) | 8 | 2
Hyponatremia (Metabolism and nutrition disorders) | 5 | 4
Radiation Mucositis (Injury, poisoning and procedural complications) | 5 | 4
Tinnitus (Ear and labyrinth disorders) | 3 | 6
Aspartate Aminotransferase Increased (Investigations) | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Fatigue (General disorders) | 2 | 6
Oral Fungal Infection (Infections and infestations) | 5 | 3
Alanine Aminotransferase Increased (Investigations) | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 4
Ear Pain (Ear and labyrinth disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 4
Pain (General disorders) | 3 | 3
Blood Bilirubin Increased (Investigations) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 2
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Edema Peripheral (General disorders) | 3 | 2
Paraesthesia (Nervous system disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Renal Failure (Renal and urinary disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Aptyalism (Gastrointestinal disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3
Epiglottic Edema (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Increased Viscosity of Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Mouth Ulceration (Gastrointestinal disorders) | 1 | 3
Oral Infection (Infections and infestations) | 2 | 2
Salivary Gland Disorder (Gastrointestinal disorders) | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1
Aphagia (Gastrointestinal disorders) | 1 | 2
Blood Sodium Decreased (Investigations) | 1 | 2
Blood Urea Increased (Investigations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 2
Chills (General disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Depressed Mood (Psychiatric disorders) | 2 | 1
Face Edema (General disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 3
Influenza (Infections and infestations) | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Neutrophil Count Increased (Investigations) | 3 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 3 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tongue Ulceration (Gastrointestinal disorders) | 0 | 3
Aphonia (Nervous system disorders) | 2 | 0
Aplasia (Congenital, familial and genetic disorders) | 2 | 0
Candidiasis (Infections and infestations) | 2 | 0
Catheter Site Infection (Infections and infestations) | 2 | 0
Depression (Psychiatric disorders) | 0 | 2
Ejection Fraction Decreased (Investigations) | 0 | 2
Fibrosis (General disorders) | 0 | 2
Gamma Glutamyltransferase Increased (Investigations) | 0 | 2
Glossitis (Gastrointestinal disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Infection (Infections and infestations) | 0 | 2
Influenza Like Illness (General disorders) | 0 | 2
Lethargy (Nervous system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 2 | 0
Rhinitis (Infections and infestations) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 2
Dental caries (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 2 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 2
White blood cell count decreased (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.